CLINICAL TRIAL: NCT03279575
Title: Testing the Efficacy of Two Behavioral Interventions at Recalibrating Physician Heuristics in Trauma Triage: a Randomized Clinical Trial
Brief Title: Testing the Efficacy of Two Behavioral Interventions at Recalibrating Physician Heuristics in Trauma Triage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Deepika Mohan, Assistant professor of critical care medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO17090094
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries | interventions — Shift Work Schedule

STUDY DESIGN:
Intervention Model Description: 1:1:1:1 allocation
Who Masked: Outcomes Assessor
Masking Description: We will mask the intervention status of participants when analyzing the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Night Shift (Experimental): Night Shift is an adventure video game with the transformational goal of teaching physicians key characteristics of patients with non-representative severe injuries - injuries classified by the American College of Surgeons as life-threatening or critical but that do not fit the archetype of injuries typically requiring treatment at a trauma center. Players take on the persona of Andy Jordan, a young emergency physician who moves home after the disappearance of his estranged grandfather (Robert Jordan) and takes up a job in the local Emergency Department (ED). In the preamble, players learn they have two explicit objectives. First, they must diagnose and treat patients who present to their ED. Second they must solve the mystery of Robert's disappearance: was he murdered or has he simply chosen to disappear?
  Interventions: Behavioral: Night Shift
- Graveyard Shift (Experimental): Graveyard Shift is a puzzle video game with the transformational goal of helping physicians derive key triage decision principles for themselves. They complete a three-step game loop to obtain case information, compare cases to determine similarities and differences between cases, and then explicitly state the decision principle that should drive decision making.
  Interventions: Behavioral: Graveyard Shift
- Educational program (Active Comparator): The educational module consists of two separate apps, both commercially available. myATLS includes a review of each chapter of the Advanced Trauma Life Support (ATLS) textbook, a series of videos demonstrating common trauma procedures, and clinical resources including checklists for use at the bedside. Trauma Life Support MCQ Review includes 550 multiple-choice questions with correct answers and explanations. The investigators will ask physicians to review the myATLS app and then com
  Interventions: Behavioral: Educational program
- Control (Placebo Comparator): Physicians in this arm will not be asked to complete any intervention.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Night Shift — Physicians in this arm of the trial will be asked to play Night Shift, an adventure video game, for two hours.
  Arms: Night Shift
Behavioral: Graveyard Shift — Physicians in this arm of the trial will be asked to play Graveyard Shift, a puzzle video game, for two hours.
  Arms: Graveyard Shift
Behavioral: Educational program — Physicians in this arm of the trial will be asked to use myATLS, an app designed by the American College of Surgeons to serve as an adjunct to the ATLS course, and Trauma Life Support MCQ Review, an app designed to help students prepare for the ATLS exam. They will be asked to spend at least two hours on the combined tasks.
  Arms: Educational program
Behavioral: Control — Physicians in this arm will serve as a no-contact control group.
  Arms: Control

SUMMARY:
The objective of this study is to compare the efficacy of two behavioral interventions at recalibrating physician heuristics.

DETAILED DESCRIPTION:
Treatment at trauma centers improves outcomes for patients with moderate-to-severe injuries. Accordingly, professional organizations, state authorities, and the federal government have endorsed the systematic triage and transfer of these patients to trauma centers either directly from the field or after evaluation at a non-trauma center. Nonetheless, between 30 to 40% of patients with moderate-to-severe injuries still only receive treatment at non-trauma centers, so-called under-triage. Most of this under-triage occurs because of physician decisions (rather than first-responder decisions). Existing efforts to change physician decision making focus primarily on knowledge of clinical practice guidelines and attitudes towards the guidelines. These strategies ignores the growing consensus that decision making reflects both knowledge as well as intuitive judgments (heuristics). Heuristics, mental short cuts based on pattern recognition, drive the majority of decision making. The investigators have developed two separate behavioral interventions to recalibrate physician heuristics in trauma triage, and will compare the effect of these interventions, an educational program, and no intervention on physician performance on a virtual simulation.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medicine physicians who work at a non-trauma center.
* Emergency medicine physicians who work at a Level III/IV trauma center.

Exclusion Criteria:

* Emergency medicine physicians who work only at a Level I/II trauma center.
* Emergency medicine physicians who do not practice in the US.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-10-29 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Incidence rate of successful triage | One month after completion of the intervention
  Physicians in all arms of the study will be asked to complete a virtual simulation, upon completion of the intervention, ideally within one month of enrollment.
  The virtual simulation replicates the environment of the ED. Physicians have to manage 10 patients that appear concurrently, while also responding to a series of audio-visual distractors. Specifically, they must provide information on whether they will admit, transfer, or discharge the patients home. The investigators will categorize severely injured patients as successfully transferred (transferred to a trauma center or died in the ED) or not (admitted). We will use a Poisson regression to estimate the association between successful transfer and exposure to the different interventions (Night Shift v. Graveyard Shift v. educational program v. control).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available on application to the investigator team.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Mohan D, Fischhoff B, Angus DC, Rosengart MR, Wallace DJ, Yealy DM, Farris C, Chang CH, Kerti S, Barnato AE. Serious games may improve physician heuristics in trauma triage. Proc Natl Acad Sci U S A. 2018 Sep 11;115(37):9204-9209. doi: 10.1073/pnas.1805450115. Epub 2018 Aug 27. PMID 30150397